CLINICAL TRIAL: NCT00019448
Title: Phase II Study of DNA Encoding the gp100 Antigen Alone or in Combination With Interleukin-2 in Patients With Recurrent Metastatic Melanoma
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066215; NCI-98-C-0086; NCT00001692 (obsolete NCT alias)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Stage IV Melanoma; Recurrent Melanoma
Keywords: adult solid tumor; body system/site cancer; cancer; melanoma; recurrent melanoma; skin tumor; solid tumor; stage IV melanoma; stage, melanoma
MeSH Terms: conditions — Melanoma; Neoplasms; Skin Neoplasms | interventions — Interleukin-2

INTERVENTIONS:
Drug: gp100 antigen
Drug: interleukin-2

SUMMARY:
RATIONALE: Vaccines made from DNA may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells. Combining vaccine therapy and interleukin-2 may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy with or without interleukin-2 in treating patients with metastatic melanoma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical response of patients receiving DNA gp100 antigen alone or in combination with interleukin-2 for recurrent metastatic melanoma.

II. Identify the immunologic response in these patients prior to and after these treatments.

III. Determine the toxicity of these treatments in these patients.

PROTOCOL OUTLINE: Patients are accrued for the first three cohorts and the study proceeds to the final two cohorts if responses are observed.

Cohort I: Patients receive gp100 antigen intramuscularly (IM) into each of 2 proximal extremities once every 4 weeks for up to 4 doses. (Closed as of December, 1999) Cohort II: Patients receive gp100 antigen intradermally (ID) at 5 sites on each of 2 proximal extremities once every 4 weeks for up to 4 doses. (Closed as of December, 1999) Cohort III: Patients receive gp100 antigen IM into each of 2 proximal extremities once every 4 weeks for up to 4 doses. If patients do not exhibit immunologic response or dose-limiting toxicity, they may receive a higher dose of gp100 antigen on subsequent courses.

Cohort IV: If cohorts I, II, or III do not produce an immune response and do not experience dose-limiting toxicity, patients receive a higher dose of gp100 antigen IM into each of 2 proximal extremities every 4 weeks for up to 4 doses.

Cohort V: Patients receive gp100 antigen IM or ID at the dose found to produce immunization once every 4 weeks for up to 4 doses. Patients also receive interleukin-2 IV over 15 minutes every 8 hours for 5 days (15 doses), beginning within 24 hours after gp100 antigen.

Patients with minor, mixed, or partial response or stable disease may receive additional courses of treatment following 3-4 weeks of rest. Patients receive a maximum of 12 courses.

Patients are followed at 4-6 weeks.

PROJECTED ACCRUAL:

A maximum of 65 patients will be accrued for this study within 1 year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Diagnosis of metastatic melanoma that has failed standard therapy Measurable disease --Prior/Concurrent Therapy-- Biologic therapy: At least 3 weeks since prior biologic therapy Chemotherapy: At least 3 weeks since prior chemotherapy Endocrine therapy: At least 3 weeks since prior endocrine therapy No concurrent steroid therapy Radiotherapy: At least 3 weeks since prior radiotherapy Surgery: Prior surgery allowed --Patient Characteristics-- Age: 16 and over Performance status: ECOG 0 or 1 Life expectancy: More than 3 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 90,000/mm3 No coagulation disorder Hepatic: Bilirubin no greater than 1.6 mg/dL ALT/AST less than 2 times normal Hepatitis B surface antigen negative Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No major cardiovascular disease Pulmonary: No major respiratory disease Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No active systemic infections No autoimmune disease No primary or secondary immunodeficiency HIV negative

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-09; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States